CLINICAL TRIAL: NCT04339920
Title: To Evaluate the Performance of a Urine Spermine Measuring Device in Predicting Prostate Biopsy Result
Brief Title: Spermine Measuring Device Evaluation Protocol
Status: Withdrawn | Type: Observational
Why Stopped: No funding
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Principal Investigator, Chinese University of Hong Kong
Other Study IDs: CRE 2020.050
Record Dates: First submitted 2020-04-02; First posted 2020-04-09 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
Keywords: Urinary spermine; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum PSA level will be collected. Up to 100cc of urine will be freshly collected from patient before they undergo prostate biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chinese patients with clinical suspicious of prostate cancer: Chinese patients with clinical suspicious of prostate cancer, due to elevated serum PSA or abnormal digital rectal examination, will be recruited for the study from the Prince of Wales Hospital and North District Hospital.
  Interventions: Diagnostic Test: Spermine Measuring Device

INTERVENTIONS:
Diagnostic Test: Spermine Measuring Device — The Spermine Measuring Device (SMD) is a simple device, with automatic urine aspiration and also spermine level assessment. First about 30 cc urine will be freshly collected by a prepared collection device. Then the cap of the SMD will be removed and the aspiration tip of the device will be immersed into the urine specimen. After firmly pressed on the device, a small sample of urine will be aspirated into the SMD. The device will then automatically assess the urine spermine level. The result will then be read at a indicator window after about 5 minutes. If the level was below a pre-set cutoff, i.e. suggestive of having increase risk of prostate cancer, the indicator window will turn into red colour. However, if the spermine level is higher than the cutoff value, i.e. low risk of having cancer, the indicator window will turn blue.

SUMMARY:
Prostate gland is a clinically important male sexual organ and its main function is for the production of semen. Globally, it is the second most common cancer in men globally and is also the fifth cancer cause for death in male. Despite the improvement in the understanding of prostate cancer, the current usage of serum prostate specific antigen (PSA) as a diagnostic marker is still not ideal. Many patients with elevated PSA and then subjected to prostate biopsy were found to have no prostate cancer. Therefore, there is a need to discover new biological markers to improve the current situation in diagnosis and also management of prostate cancer. In our recent studies, urinary spermine levels have been shown to correlate well with prostate cancer diagnosis and cancer aggressiveness.

Due to its nature, it could provide a more convenient and non-invasive method for detecting prostate cancer. In order to further improve the accessibility of the test, a simple urine measuring device has been designed to allow more simple and practical usage of the test in clinical setting.The purpose of this study was to evaluate the accuracy of this newly designed urine measuring device for urinary spermine in predicting your prostatic biopsy result.

DETAILED DESCRIPTION:
Prostate cancer (PC) is highly prevalent worldwide and is currently the 3rd most commonly diagnosed prostate cancer in Hong Kong male population with more than 2000 new cases diagnosed per year. Depending on the clinical staging and also the patients' condition, different treatments, including curative surgery or radiotherapy, palliative androgen deprivation therapy, could be offered to patients and will good response. However, current there are only one biological marker, PSA, for the monitoring of the disease progress and treatment response. While PSA testing provided a reasonable assessment of the disease status and progress, it is an invasive blood test and maybe less convenience for some patients. Therefore, there is a need for exploring newer markers for the monitoring of the treatment response and disease progress is needed.

One example of such cancer biomarkers are natural polyamines. Interests on these analytes have been starting in 1971 when Russell reported a considerable increase of urinary polyamines such as putrescine (Put), spermidine (Spd) and spermine (Spm) in patients with various types of solid tumors and leukaemias. Afterwards, polyamine studies focusing on specific cancers continued, like cervical cancer, colorectal cancer and breast cancer, etc.

In our recent study, we have explored the potential roles of urinary polyamines as prostate cancer biomarkers were evaluated. Patients with prostate cancer (PCa), benign prostatic hyperplasia (BPH) patients and healthy controls (HC) showing PSA>4.0ng/ml were enrolled in the study. Their urine samples were obtained, and the urinary levels of Put, Spd, Spm were determined by ultra-high-performance liquid chromatography coupled with triple quadrupole mass spectrometer (UPLC-MS/MS). Receiver operating characteristics (ROC) curve and Student's t- test were used to evaluate their diagnostic accuracies. Among the three biogenic polyamines, Spm had demonstrated a good diagnostic performance when comparing their levels in PCa patients with BPH patients (1.47 in PCa vs 5.87 in BPH; p<0.0001). The results were in accordance with transrectal ultrasound prostatic biopsy (TRUSPB) results, with an area under curve (AUC) value of 0.83±0.03. Therefore, urinary Spm could have a potential to serve as a novel PCa diagnostic biomarker, which in turn could help to address the limited sensitivity and specificity problem of serum PSA test. In our further work, we have confirmed that spermine is a good marker for the detection of prostate cancer and also showed good correlation with cancer grading.

However, the current measurement of spermine required the use of liquid chromatography (LCM) in laboratory, which might limit its clinical usage. Therefore, a simple spermine measuring device (SMD) has been designed for easier daily usage, such as simple cancer screening and also combined evaluation with serum PSA level. The SMD is a simple device, with automatic urine aspiration and also spermine level assessment. First about 30 cc urine will be freshly collected by a prepared collection device. Then the cap of the SMD will be removed and the aspiration tip of the device will be immersed into the urine specimen. After firmly pressed on the device, a small sample of urine will be aspirated into the SMD. The device will then automatically assess the urine spermine level. The result will then be read at a indicator window after about 5 minutes. If the level was below a pre-set cutoff, i.e. suggestive of having increase risk of prostate cancer, the indicator window will turn into red colour.

However, if the spermine level is higher than the cutoff value, i.e. low risk of having cancer, the indicator window will turn blue. However, the kit has not been validated in clinical urine sample. Therefore, we would like to perform an evaluation the accuracy of this SMD with the laboratory measured spermine level by LCM, as well as the pathology result from prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Adult Chinese male patients with age > 18 years old
* Clinical indicated for prostate cancer detection and has serum PSA level done within 8 weeks of urine test.

Exclusion Criteria:

* Patient with recent urinary tract infection within 6 weeks prior to urine collection.
* Patient with recent urethral instrumentation, such as Foley catheter insertion, cystoscopy etc., within 6 weeks prior to urine collection.
* Patient with consumption of 5 alpha reductase inhibitors in past 6 months.
* Patient refused or unable to provide consent for the study

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate can only be found in male
Study Population: Chinese patients with clinical suspicious of prostate cancer, due to elevated serum PSA or abnormal digital rectal examination, will be recruited for the study from the Prince of Wales Hospital and North District Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Correlation of the Spermine measuring device and final prostate biopsy results. | At baseline
  By comparing the urine spermine level results of the spermine measuring device with the prostate biopsy pathology

SECONDARY OUTCOMES:
Accuracy of the Spermine measuring device in measuring the urine spermine level | At baseline
  By comparing the urine spermine level results of the spermine measuring device with that of the liquid chromatography

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Hong Kong Cancer registry 2017.
- [Background] Wong HF, Yee CH, Teoh JY, Chan SY, Chiu PK, Cheung HY, Hou SS, Ng CF. Time trend and characteristics of prostate cancer diagnosed in Hong Kong (China) in the past two decades. Asian J Androl. 2019 Jan 1;21(1):104-106. doi: 10.4103/aja.aja_75_18. No abstract available. PMID 30178778
- [Background] Russell DH. Increased polyamine concentrations in the urine of human cancer patients. Nat New Biol. 1971 Sep 29;233(39):144-5. doi: 10.1038/newbio233144a0. No abstract available. PMID 5286749
- [Background] Lee SH, Yang YJ, Kim KM, Chung BC. Altered urinary profiles of polyamines and endogenous steroids in patients with benign cervical disease and cervical cancer. Cancer Lett. 2003 Nov 25;201(2):121-31. doi: 10.1016/s0304-3835(03)00014-4. PMID 14607325
- [Background] Loser C, Folsch UR, Paprotny C, Creutzfeldt W. Polyamines in colorectal cancer. Evaluation of polyamine concentrations in the colon tissue, serum, and urine of 50 patients with colorectal cancer. Cancer. 1990 Feb 15;65(4):958-66. doi: 10.1002/1097-0142(19900215)65:43.0.co;2-z. PMID 2297664
- [Background] Leveque J, Foucher F, Bansard JY, Havouis R, Grall JY, Moulinoux JP. Polyamine profiles in tumor, normal tissue of the homologous breast, blood, and urine of breast cancer sufferers. Breast Cancer Res Treat. 2000 Mar;60(2):99-105. doi: 10.1023/a:1006319818530. PMID 10845272
- [Background] Tsoi TH, Chan CF, Chan WL, Chiu KF, Wong WT, Ng CF, Wong KL. Urinary Polyamines: A Pilot Study on Their Roles as Prostate Cancer Detection Biomarkers. PLoS One. 2016 Sep 6;11(9):e0162217. doi: 10.1371/journal.pone.0162217. eCollection 2016. PMID 27598335
- [Background] Chiu PKF, Tsoi TH, Wong YP, Teoh JYC, Lo KL, Ng CF, Wong KL. The novel urine Spermine test predicts prostate cancer: the first prospective evaluation. (Accepted poster presentation in EAU 2020)